CLINICAL TRIAL: NCT06682975
Title: A First-in-human, Randomized and Double-blind Within Cohorts, Placebo-controlled, Single Ascending Dose Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZP9830 Administered to Healthy Male Subjects.
Brief Title: A Research Study Looking at the Safety of Single Doses of ZP9830 and How it Works in the Body of Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ZP9830-23005; 2023-509929-51-00 (EU CTIS Number); 2023-509929-51 (EudraCT Number); U1111-1305-8892 (Other: World Health Organisation, WHO, UTN number)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Parallel (active or placebo), sequential (dose escalation)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZP9830 (Experimental): Up to 10 single cohorts planned:
  Part A, 3 cohorts of each 8 participants with 6 participants receiving s.c. active treatment of ZP9830. Part B, 6 cohorts of each 10 participants with 8 participants receiving s.c. active treatment of ZP9830. Part C, 1 cohort of 8 participants with 6 participants receiving i.v. active treatment of ZP9830
  Interventions: Drug: ZP9830
- Placebo (Placebo Comparator): In each of the 10 single dose cohorts, 2 subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZP9830 — Participants will receive 1 single dose of ZP9830 given subcutaneously (s.c., under the skin) or intravenously (i.v., in a vein of the arm). Dose level will depend on the cohort.
  Arms: ZP9830
Drug: Placebo — Participants will receive 1 single dose of placebo given subcutaneously (s.c., under the skin) or intravenously (i.v., in a vein of the arm). Volume will be matching the active treatment
  Arms: Placebo

SUMMARY:
The primary object in this research study is to investigate the safety and tolerability of ZP9830 in healthy study participants, and in addition, the study will investigate how ZP9830 works in the body (pharmacokinetics, PK and pharmacodynamics, PD) compared to placebo.

DETAILED DESCRIPTION:
Part A: Participants will receive 1 dose either ZP9830 or placebo as an injection under the skin (subcutaneous, s.c), and safety and PK will be assessed.

Part B: Participants will receive 1 dose either ZP9830 or placebo as an injection under the skin (subcutaneous, s.c.) and safety, PK and PD will be assessed.

Part C: Participants will receive 1 dose either ZP9830 or placebo as intravenous (i.v.) dose, and safety and PK will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Healthy male subject.

18-45 years of age (inclusive).

Body weight ≥50 kg.

Part B only: Fitzpatrick skin type I-III (Caucasian).

C-reactive protein ≤10 mg/L.

Further inclusion criteria apply.

Exclusion Criteria:

Evidence of any active or chronic disease or condition that could interfere with, or for which the treatment of it might interfere with, the conduct or the interpretation of the results of the trial, or that would pose an unacceptable risk to the subject in the opinion of the Investigator [following a detailed medical history, physical examination, vital signs (systolic and diastolic blood pressure, pulse rate, body temperature) and 12-lead ECG].

Any disease associated with immune system impairment, including immune mediated diseases and transplantation patients.

Any confirmed significant allergic reactions (urticaria or anaphylaxis) to insect bites.

History of neurological disorders including neuropathy, as judged by the investigator.

Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug or food (in particular any level of severity of allergy to shellfish), or multiple drug allergies (non-active hay fever is acceptable).

Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incident of Treatment Emergent Adverse Events (TEAEs) | From dosing of ZP9830 (Day 1) to follow-up (Day 29)
  Treatment Emergent Adverse Events (TEAEs) from baseline to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zealand Pharma A/S, Study Director — Zealand Pharma A/S
Locations (1):
- Centre for Human Drug Research, Leiden, CL, Netherlands

IPD SHARING:
Plan to Share IPD: No